CLINICAL TRIAL: NCT05500040
Title: Veränderungen Des Faecalen Calprotectinwertes Und Teilhabebezogener Scores in Folge Einer Dreiwöchigen Phase II Rehabilitation [Changes in Faecal Calprotectin Levels and Participation-related Scores Following Three Weeks of Inpatient Rehabilitation]
Brief Title: Changes in Faecal Calprotectin Levels and Participation-related Scores Following Three Weeks of Inpatient Rehabilitation
Status: Completed | Type: Observational
Sponsor: Pensionsversicherungsanstalt (Other)
Responsible Party: Sponsor
Other Study IDs: 0008-CED
Record Dates: First submitted 2022-08-09; First posted 2022-08-12 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-01

CONDITIONS: Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with IBD - Crohn's Disease
  Interventions: Behavioral: Multimodal Rehabilitation
- Patients with IBD - Ulcerative Colitis
  Interventions: Behavioral: Multimodal Rehabilitation

INTERVENTIONS:
Behavioral: Multimodal Rehabilitation — The rehabilitation measure is based on the biopsychosocial ICF model of the WHO. A multidisciplinary team of therapists looks after the patients during their stay in rehabilitation. Taking into account the physical and psychological condition of the patients, an individual therapy plan is created that is tailored to their needs.

SUMMARY:
For many people affected by inflammatory bowel disease (IBD), their quality of life and their ability to participate in their professional and social lives are severely restricted. Rehabilitation measures based on the biopsychosocial ICF model aim to support the restoration of these abilities. Physiological parameters (e.g. biomarkers) as well as patient-reported outcomes (PROs) can be used to assess the success of ICF-based rehabilitation measures and to optimize them. A suitable biomarker to monitor inflammation in IBD patients is faecal calprotectin. In addition, PROs that support patients in providing information, for example on their health-related quality of life or on their subjective ability to work, can provide information on the individual social and occupational participation ability of the patients. The aim of this project is to investigate changes in a biomarker (calprotectin) as well as in selected PROs after a three-week inpatient phase II rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Crohn's Disease or Ulcerative Colitis
* Participation in an inpatient phase II rehabilitation

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Rehabilitation patients with IBD in inpatient rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Faecal Calprotectin | 3 weeks of inpatient rehabilitation
  Faecal calprotectin is a biochemical measurement of the protein calprotectin in the stool. Elevated faecal calprotectin indicates the migration of neutrophils to the intestinal mucosa, which occurs during intestinal inflammation, including inflammation caused by inflammatory bowel disease.
Ced Disk | 3 weeks of inpatient rehabilitation
  The Ced Disk measures IBD-related impairments in different dimensions i.e., abdominal pain, bowel control, interpersonal interactions, education and work, sleep, energy, emotions, body image, sexuality, joint pain (Min. = 0, Max. = 10). Lower values indicate less impairments in the respective dimensions.
European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) | 3 weeks of inpatient rehabilitation
  The EQ-5D-5L is a general instrument for measuring patient-reported outcomes (PROs), which can be used to assess the quality of life of patients on different dimensions (mobility, self-care, usual activities, pain/discomfort) on a 5-level scale (Min. = 0, Max. = 5). Lower values indicate less impairments in the respective dimensions.
  Moreover, the EQ-5D-5L assesses the patient's self-rated health on a 100 point visual analog scale (Min. = 0, Max. = 100). Lower values indicate less positive ratings of health.
Patient Health Questionnaire-4 (PHQ-4) | 3 weeks of inpatient rehabilitation
  The Patient Health Questionnaire-4 (PHQ-4) operationalizes core criteria for anxiety and depression on a 4 point likert scale (Min. = 0, Max = 4). Lower values indicate less impairments.
Work ability index (WAI) | 3 weeks of inpatient rehabilitation
  The Work Ability Index (WAI) is an instrument for assessing work ability. (Min. = 7, Max = 49). Lower values indicate less subjective work ability.

CONTACTS AND LOCATIONS:
Overall Officials: Doreen Stöhr, Mag., Study Chair — Pensionsversicherungsanstalt
Locations (1):
- Rehabilitationszentrum Bad Aussee, Vienna, Styria, Austria

IPD SHARING:
Plan to Share IPD: No